CLINICAL TRIAL: NCT05813431
Title: Randomized Controlled Pilot Study of Methods for Identifying Patients At High Risk of Worsening in the Adult Emergency Department
Acronym: Quick-TRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GALOPIN AOIparaM 2021
Record Dates: First submitted 2023-04-03; First posted 2023-04-14 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Non-traumatic Medical Emergency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control - FRENCH grid only (Active Comparator)
  Interventions: Other: FRENCH grid (classification for emergency nurses in French hospitals)
- FRENCH grid + QuickSOFA (Active Comparator)
  Interventions: Other: FRENCH grid (classification for emergency nurses in French hospitals); Other: QuickSOFA
- FRENCH grid + QuickSOFA + Capillary Lactate (Active Comparator)
  Interventions: Other: FRENCH grid (classification for emergency nurses in French hospitals); Other: QuickSOFA; Other: Capillary lactate assessment

INTERVENTIONS:
Other: FRENCH grid (classification for emergency nurses in French hospitals) — Triage tool validated by the French Society of Emergency Medicine (SFMU) which is used to prioritize patients according to standardized criteria and to orient them within the emergency department.
Other: QuickSOFA — Rapid score that consists of an evaluation based on 3 clinical criteria (blood pressure, respiratory rate and consciousness) to quickly establish a severity score.
  Arms: FRENCH grid + QuickSOFA; FRENCH grid + QuickSOFA + Capillary Lactate
Other: Capillary lactate assessment — Collect a drop of blood from the fingertip (less than 1 ml)
  Arms: FRENCH grid + QuickSOFA + Capillary Lactate

SUMMARY:
This study will be conducted in the Regional Emergency Room (ER) of the Dijon-Bourgogne University Hospital in Dijon, France. It is an interventional study that will have an impact on medical contact time.

Patients will be identified among adult patients presenting to the ER of the Dijon University Hospital. Each patient will be followed-up for 30 days from the time of arrival at the ER (if the inclusion criteria for the study are met).

A total of 337 patients will participate in this study and will be randomly allocated to 3 groups:

* Group 1 "controls - FRENCH grid only": patients will receive the same care and management as any other patient admitted for the same condition. Management is based on the use of the FRENCH grid only.
* Group 2 "FRENCH grid + QuickSOFA": In addition to the standard use of the FRENCH grid, a quick score called QuickSOFA is added. It consists in performing an evaluation based on 3 clinical criteria (blood pressure, respiratory rate and consciousness) to quickly establish a severity score.
* Group 3 "FRENCH grid + QuickSOFA + Capillary lactate": In addition to the use of the FRENCH grid and the QuickSOFA score, capillary lactate concentrations will be measured. This involves taking a drop of blood from the fingertip (less than 1ml). For diabetic patients, there will be no second sampling act, everything will be done from the same sample. All samples will be discarded after the result is displayed on the reader.

This study includes 2 visits:

- D0 (adult ER visit): The patient's background, clinical and biological data will be collected. The patient will then be randomized into one of three groups. Depending on the group assigned, the triage nurse may perform QuickSOFA and lactate assessments.

- Follow-up at D30: collection of follow-up information up to 30 days after inclusion in the emergency department: replacement therapy (mechanical ventilation, extracorporeal membrane oxygenation,…), dates of discharge from critical care and hospital, vital status and in case of death the date of its occurrence.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients admitted to the Dijon-Bourgogne University Hospital emergency room between 12:00 am and 10:00 pm on weekdays for a medical emergency (non-traumatic)
* Patients classified 3A 3B according to the FRENCH triage grid
* Patient who gives verbal informed consent to take part in the study
* Patient affiliated with national healthcare coverage (if not, the patient is redirected to the permanence of access to health care - PASS).

Exclusion Criteria:

* Patients admitted to the ER by the emergency services or having had a complete check-up in relation to the reason for transfer to the ER, therefore having had medical contact before hospital admission
* Patients under palliative care for a defined condition
* Person under legal protection (curatorship, guardianship)
* Person under court order
* Pregnant, parturient or breastfeeding woman
* Adult who is unable to express consent

Secondary exclusion criteria:

- Patients admitted for a stroke or suspected stroke referred either directly or after a delay to the specific stroke care pathway are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 337 (Actual)
Dates: Start 2023-09-08 (Actual); Primary Completion 2024-12-27 (Actual); Study Completion 2024-12-27 (Actual)

PRIMARY OUTCOMES:
Waiting time in minutes between contact with the triage nurse and the first medical contact in the emergency room | At inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France

IPD SHARING:
Plan to Share IPD: No